CLINICAL TRIAL: NCT00416871
Title: Cytokines in the Treatment of Metastatic Renal Cell Carcinoma (MRCC): Intravenous Interleukin and Subcutaneous Interferon-α Versus Subcutaneous Interleukin and Interferon-α for Good Prognosis Patients [PERCY DUO]
Brief Title: Interleukin-2 and Interferon in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000468028; LEONB-PERCY-DUO; LEONB-ET99-057; EU-20604; ROCHE-LEONB-PERCY-DUO; CHIRON-LEONB-PERCY-DUO
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin; Interferon-alpha

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon alfa

SUMMARY:
RATIONALE: Biological therapies, such as interleukin-2 and interferon, may stimulate the immune system in different ways and stop tumor cells from growing. It is not yet known whether interleukin-2 given by infusion is more effective than interleukin-2 given by injection when combined with interferon in treating metastatic kidney cancer.

PURPOSE: This randomized phase III trial is studying interleukin-2 given by infusion to see how well it works compared to interleukin-2 given by injection when combined with interferon in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with metastatic renal cell cancer treated with intravenous vs subcutaneous interleukin-2 in combination with interferon alfa.

Secondary

* Compare progression-free survival of patients treated with these regimens.
* Compare response rates (complete and partial) in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare quality of life of patients treated with these regimens.

OUTLINE: This is an open-label, randomized, parallel-group, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive induction therapy comprising interleukin-2 (IL-2) IV continuously over days 1-5, 15-19, 43-47, and 57-61 (weeks 1, 3, 7, and 9) and interferon alfa (IFN-α) subcutaneously (SC) three times weekly in weeks 1-3 and 7-9. Patients then undergo restaging. Patients achieving a complete response (CR), partial response (PR), or stable disease (SD) then receive maintenance therapy comprising IL-2 IV continuously over 5 days and IFN-α SC three times weekly in weeks 1, 5, 9, and 13.
* Arm II: Patients receive induction therapy comprising IL-2 SC twice daily on days 1-5, 8-12, 15-19, and 22-26 (weeks 1-4). Patients also receive IFN-α SC three times weekly in weeks 1-4 and 6-9. Patients then undergo restaging. Patients achieving a CR, PR, or SD then receive maintenance therapy comprising IL-2 SC as in induction therapy and IFN-α SC three times weekly in weeks 1-4 and 8-11.

Quality of life is assessed at baseline, at the end of induction therapy, and then at the end of maintenance therapy.

After completion of treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 220 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic renal cell adenocarcinoma

  * More than one resectable metastatic site
  * No unresectable lesions after local curative treatment (i.e., radiotherapy)
  * In case of secondary lesions suspected on imaging (< 1 cm and/or sparse lesions), metastatic disease must be confirmed by biopsy OR disease progression documented by imaging performed over several weeks
  * If patient has known prior metastatic lesions, progressive disease must have been confirmed within the past 3 months by noninvasive techniques
* Nephrectomized
* Measurable or evaluable disease
* No brain metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status 90-100%
* Hematocrit ≥ 30%
* WBC ≥ 4,000/mm^3
* Platelet count ≥ 120,000/mm^3
* Bilirubin normal
* Creatinine ≤ 1.7 mg/dL
* FEV_1 ≥ 50%
* No severe cardiac dysfunction (i.e., grade III/IV heart disease), including any of the following:

  * Congestive heart failure
  * Coronary artery disease
  * Uncontrolled hypertension
  * Severe arrhythmia
* No active infections requiring antibiotic treatment
* No severe neuropsychiatric condition
* No geographical, psychological, or familial conditions that would preclude study treatment
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* LVEF ≥ 50%
* No severe autoimmune disease
* No known chronic hepatitis
* No HIV positivity
* No hepatitis B surface antigen positivity
* No prior or concurrent other cancer, except basal cell skin cancer or carcinoma in situ of the cervix
* No severe pulmonary, hepatic, or renal condition that would preclude study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 6 weeks since prior wide-field radiotherapy
* No prior allograft
* No prior cytokines or chemotherapy
* No concurrent corticosteroids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Negrier, MD, Study Chair — Centre Leon Berard

REFERENCES:
- [Result] Negrier S, Perol D, Ravaud A, Bay JO, Oudard S, Chabaud S, Fargeot P, Delva R, Deplanque G, Gravis G, Escudier B; French Immunotherapy Group. Randomized study of intravenous versus subcutaneous interleukin-2, and IFNalpha in patients with good prognosis metastatic renal cancer. Clin Cancer Res. 2008 Sep 15;14(18):5907-12. doi: 10.1158/1078-0432.CCR-08-0236. PMID 18794104